CLINICAL TRIAL: NCT03133338
Title: Division of Traumatic and General Surgery, Department of Surgery, Tri-Service General Hospital, National Defense Medical Center
Brief Title: Effect of Early Pelvic Binder Use in Emergency Management of Suspected Pelvic Trauma: a Retrospective Cohort Study
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Hsu Sheng-Der, Division of Traumatic and General Surgery, Department of Surgery, Tri-Service General Hospital, National Defense Medical Center, Tri-Service General Hospital
Other Study IDs: TSGHIRB No. 1-103-05-122
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Fracture
MeSH Terms: conditions — Hip Fractures | interventions — Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: pelvic binder — The requirement of angioembolization can be predicted by the presence of intravenous contrast extravasation (ICE) on computed tomography (CT)
  Other Names: Angiography for TAE

SUMMARY:
The investigators aimed to evaluate the effect of early pelvic binder use in emergency management of suspected pelvic trauma, compared with the conventional stepwise approach.

DETAILED DESCRIPTION:
There is currently no universal consensus on all aspects of management of pelvic injuries.

Among patients with multiple injuries because of blunt trauma, 5%-16% sustain injuries to the pelvic ring, resulting in a mortality rate of 11%-54% primarily due to hemorrhagic shock. In theory, the reduction and stabilization of the pelvic ring can decrease bleeding from the fracture site, as reduction of pelvic volume has been shown to reduce the extent of hemorrhage from such injuries.The application of a pelvic binder has become part of the emergency care of all trauma patients with suspected pelvic fractures, in both the pre-hospital environment and emergency department (ED). The present study aimed to assess the effectiveness of the early use of pelvic binders to treat patients with a suspected high risk of pelvic bleeding from blunt force pelvic fractures.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic injury requiring a trauma team and at least one of the following: loss of consciousness or Glasgow coma score (GCS) < 13; systolic blood pressure < 90 mmHg; falling from ≥6 m; injury to multiple vital organs; and suspected pelvic injury. -

Exclusion Criteria:

* Not meet the criteria and loss follow up (transfer to other hospital or data not available) -

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We enrolled trauma patients with initial stabilization using a pelvic binder for suspecting pelvic injury. Inclusion criteria were traumatic injury requiring a trauma team and at least one of the following: loss of consciousness or Glasgow coma score (GCS) < 13; systolic blood pressure < 90 mmHg; falling from ≥6 m; injury to multiple vital organs; and suspected pelvic injury. Various parameters, including gender, age, mechanism of injury, GCS, mortality, hospital stay, initial vital sign, revised trauma score, injury severity score, and outcome, were assessed and compared with historical controls.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-07-31 (Actual); Study Completion 2014-07-31 (Actual)

PRIMARY OUTCOMES:
Blood transfusion | admission
  Pelvic fracture with hemodynamic unstable

SECONDARY OUTCOMES:
admission mortality | mortality in the same admission
  mortality in the same admission

CONTACTS AND LOCATIONS:
Overall Officials: Mu-Hsien Yu, Professor, Study Director — Institutional Review Board II of the Tri-Service General Hospital, National Defense Medical Center.